CLINICAL TRIAL: NCT04906499
Title: Preventing Posttraumatic Osteoarthritis With Physical Activity Promotion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-0614; 2KR1372103 (Other Grant/Funding Number: North Carolina Translational and Clinical Sciences Institute)
Record Dates: First submitted 2021-05-25; First posted 2021-05-28 (Actual); Results first posted 2024-01-29 (Actual); Last update posted 2024-01-29 (Actual); Status verified 2023-04

CONDITIONS: Anterior Cruciate Ligament Injuries; Exercise; Cartilage, Articular; Knee Injuries; Osteoarthritis; Osteoarthritis, Knee; Arthritis; Joint Diseases
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Motor Activity; Knee Injuries; Osteoarthritis; Osteoarthritis, Knee; Arthritis; Joint Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physical Activity Promotion Group (Experimental): Participants will receive a text message each morning with a personalized, daily step count goal and a link used to confirm receipt of the goal. The preceding 10 days of step data will be rank ordered and the 60th percentile step count will be set as the goal for the next day.
  Interventions: Behavioral: Physical Activity Promotion

INTERVENTIONS:
Behavioral: Physical Activity Promotion — After enrolling, participants will be outfitted with a Fitbit Charge 2 activity monitor. The monitor will be worn during all waking hours, and compliance will be considered as a day with ≥ 1,000 steps. Participants will complete a 14-day "run-in" observation period while wearing the Fitbit but no PA promotion will occur. Individuals who are noncompliant during the "run in" period (<10 days with <1,000 steps) will be removed. Participants will receive a text message each morning with a personalized, daily step count goal and a link used to confirm receipt of the goal. The preceding 10 days of step data will be rank ordered and the 60th percentile step count will be set as the goal for the next day.

SUMMARY:
Osteoarthritis (OA) is a leading cause of disability worldwide that affects millions of Americans each year. Posttraumatic OA (PTOA) significantly impacts patients after anterior cruciate ligament (ACL) injury and ACL reconstruction (ACLR) with approximately 50% of patients developing PTOA within 20 years of injury or surgery. Knee joint mechanical loading measured via physical activity (i.e. daily steps) is insufficient in individuals after ACLR compared to uninjured individuals. Establishing the beneficial effects of physical activity to promote optimal free-living knee joint mechanical loading and improve knee joint health will aid in the development of cost-effective interventions that prevent PTOA and health burden of the disease.

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a leading cause of disability worldwide resulting in severe limitations in daily activities and chronic pain. It is estimated that 35% of posttraumatic OA (PTOA) cases occur after knee injuries and surgeries such as anterior cruciate ligament (ACL) injury and ACL reconstruction (ACLR). Optimal free-living mechanical loading, which refers to the forces acting on the knee caused by daily activities, plays an essential role in maintaining knee articular cartilage health. After ACLR, individuals take fewer steps per day as compared to uninjured controls. This results in insufficient free-living mechanical loading to joint tissues and is associated with early PTOA development. Adequate physical activity (PA) is recommended to help reduce risk of PTOA, but it is unclear how changes in PA acutely impact knee joint cartilage health. The overall objective of this pretest-posttest experimental pilot study is to determine how optimizing free-living mechanical loading through PA promotion improves cartilage composition in individuals who demonstrate insufficient free-living mechanical loading after ACLR. PA promotion will be delivered over 8 weeks using commercially available PA monitors and the patients' smartphone to provide daily personalized and achievable step goals to increase daily step counts to a level consistent with healthy PA participation. The hypothesis for aim 1 is that MRI markers of proteoglycan density associated with PTOA development will improve after 8-weeks of PA promotion exposure. Hypothesis for aim 2 is that greater changes in steps per day will be associated with improved proteoglycan density. Change in MRI markers of proteoglycan density and steps per day will be assessed using a pretest-posttest design in 8 adults who are 6 months to 5 years post-ACLR with insufficient mechanical loading (<8,000 steps per day)24 and suboptimal quality of life (quality of life survey<87.5). Outcomes will be collected before (pretest) and after (posttest) 8-weeks of PA promotion. For the PA promotion, participants will receive a text message each morning with a personalized, daily step count goal and a link used to confirm receipt of the goal. The preceding 10 days of step data will be rank ordered and the 60th percentile step count will be set as the goal for the next day. The proposed work is innovative, in that this study will use a novel combination of outcomes that will lead to unprecedented insight into the influence of PA promotion in mitigating early PTOA development.

ELIGIBILITY:
Inclusion Criteria

Participants will be included if they:

* Provide informed consent and sign a HIPPA form prior to any study procedures are performed
* Have completed all other formal physical therapy and therapeutic exercise regimens, and will not be engaging in any other formal therapy for their ACLR during the study
* Are between the ages of 18 and 35.
* Underwent an ACLR no earlier than 6 months and no later than 5 years prior to enrollment.
* Demonstrate < 8,000 steps per day during the screening phase of the study as assessed using the Actigraph GT9X Link monitor.
* Demonstrate clinically relevant-knee symptoms, defined as a Knee Injury and Osteoarthritis Outcomes Score (KOOS) quality of life subscale < 72.2

Exclusion Criteria

Participants will be excluded if:

* The participant underwent an ACLR revision surgery due to a previous ACL graft injury.
* Multiple ligament surgery was indicated at the time of ACLR surgery.
* A lower extremity fracture was suffered during the ACL injury.
* The participant has been diagnosed with osteoarthritis in either knee
* They have a cochlear implant, metal in body, claustrophobia, or history of seizures.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Pietrosimone, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Fetzer Hall, University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Time Frame: 9 to 36 months
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.

REFERENCES:
- [Background] Cross M, Smith E, Hoy D, Nolte S, Ackerman I, Fransen M, Bridgett L, Williams S, Guillemin F, Hill CL, Laslett LL, Jones G, Cicuttini F, Osborne R, Vos T, Buchbinder R, Woolf A, March L. The global burden of hip and knee osteoarthritis: estimates from the global burden of disease 2010 study. Ann Rheum Dis. 2014 Jul;73(7):1323-30. doi: 10.1136/annrheumdis-2013-204763. Epub 2014 Feb 19. PMID 24553908
- [Background] Lawrence RC, Felson DT, Helmick CG, Arnold LM, Choi H, Deyo RA, Gabriel S, Hirsch R, Hochberg MC, Hunder GG, Jordan JM, Katz JN, Kremers HM, Wolfe F; National Arthritis Data Workgroup. Estimates of the prevalence of arthritis and other rheumatic conditions in the United States. Part II. Arthritis Rheum. 2008 Jan;58(1):26-35. doi: 10.1002/art.23176. PMID 18163497
- [Background] Furner SE, Hootman JM, Helmick CG, Bolen J, Zack MM. Health-related quality of life of US adults with arthritis: analysis of data from the behavioral risk factor surveillance system, 2003, 2005, and 2007. Arthritis Care Res (Hoboken). 2011 Jun;63(6):788-99. doi: 10.1002/acr.20430. PMID 21538946
- [Background] Alkan BM, Fidan F, Tosun A, Ardicoglu O. Quality of life and self-reported disability in patients with knee osteoarthritis. Mod Rheumatol. 2014 Jan;24(1):166-71. doi: 10.3109/14397595.2013.854046. PMID 24261774
- [Background] Brown TD, Johnston RC, Saltzman CL, Marsh JL, Buckwalter JA. Posttraumatic osteoarthritis: a first estimate of incidence, prevalence, and burden of disease. J Orthop Trauma. 2006 Nov-Dec;20(10):739-44. doi: 10.1097/01.bot.0000246468.80635.ef. PMID 17106388
- [Background] Luc B, Gribble PA, Pietrosimone BG. Osteoarthritis prevalence following anterior cruciate ligament reconstruction: a systematic review and numbers-needed-to-treat analysis. J Athl Train. 2014 Nov-Dec;49(6):806-19. doi: 10.4085/1062-6050-49.3.35. PMID 25232663
- [Background] Murphy L, Schwartz TA, Helmick CG, Renner JB, Tudor G, Koch G, Dragomir A, Kalsbeek WD, Luta G, Jordan JM. Lifetime risk of symptomatic knee osteoarthritis. Arthritis Rheum. 2008 Sep 15;59(9):1207-13. doi: 10.1002/art.24021. PMID 18759314
- [Background] Andriacchi TP, Mundermann A. The role of ambulatory mechanics in the initiation and progression of knee osteoarthritis. Curr Opin Rheumatol. 2006 Sep;18(5):514-8. doi: 10.1097/01.bor.0000240365.16842.4e. PMID 16896293
- [Background] Bell DR, Pfeiffer KA, Cadmus-Bertram LA, Trigsted SM, Kelly A, Post EG, Hart JM, Cook DB, Dunn WR, Kuenze C. Objectively Measured Physical Activity in Patients After Anterior Cruciate Ligament Reconstruction. Am J Sports Med. 2017 Jul;45(8):1893-1900. doi: 10.1177/0363546517698940. Epub 2017 Apr 18. PMID 28419817
- [Background] Nelson AE, Allen KD, Golightly YM, Goode AP, Jordan JM. A systematic review of recommendations and guidelines for the management of osteoarthritis: The chronic osteoarthritis management initiative of the U.S. bone and joint initiative. Semin Arthritis Rheum. 2014 Jun;43(6):701-12. doi: 10.1016/j.semarthrit.2013.11.012. Epub 2013 Dec 4. PMID 24387819
- [Background] Palmieri-Smith RM, Cameron KL, DiStefano LJ, Driban JB, Pietrosimone B, Thomas AC, Tourville TW, Consortium ATO. The Role of Athletic Trainers in Preventing and Managing Posttraumatic Osteoarthritis in Physically Active Populations: a Consensus Statement of the Athletic Trainers' Osteoarthritis Consortium. J Athl Train. 2017 Jun 2;52(6):610-623. doi: 10.4085/1062-6050-52.2.04. PMID 28653866
- [Background] Tudor-Locke C, Craig CL, Brown WJ, Clemes SA, De Cocker K, Giles-Corti B, Hatano Y, Inoue S, Matsudo SM, Mutrie N, Oppert JM, Rowe DA, Schmidt MD, Schofield GM, Spence JC, Teixeira PJ, Tully MA, Blair SN. How many steps/day are enough? For adults. Int J Behav Nutr Phys Act. 2011 Jul 28;8:79. doi: 10.1186/1479-5868-8-79. PMID 21798015
- [Background] Ingelsrud LH, Granan LP, Terwee CB, Engebretsen L, Roos EM. Proportion of Patients Reporting Acceptable Symptoms or Treatment Failure and Their Associated KOOS Values at 6 to 24 Months After Anterior Cruciate Ligament Reconstruction: A Study From the Norwegian Knee Ligament Registry. Am J Sports Med. 2015 Aug;43(8):1902-7. doi: 10.1177/0363546515584041. Epub 2015 May 14. PMID 25977523
- [Background] Roos EM, Toksvig-Larsen S. Knee injury and Osteoarthritis Outcome Score (KOOS) - validation and comparison to the WOMAC in total knee replacement. Health Qual Life Outcomes. 2003 May 25;1:17. doi: 10.1186/1477-7525-1-17. PMID 12801417
- [Background] Pfeiffer S, Harkey MS, Stanley LE, Blackburn JT, Padua DA, Spang JT, Marshall SW, Jordan JM, Schmitz R, Nissman D, Pietrosimone B. Associations Between Slower Walking Speed and T1rho Magnetic Resonance Imaging of Femoral Cartilage Following Anterior Cruciate Ligament Reconstruction. Arthritis Care Res (Hoboken). 2018 Aug;70(8):1132-1140. doi: 10.1002/acr.23477. Epub 2018 Jul 4. PMID 29193888
- [Background] Pietrosimone B, Nissman D, Padua DA, Blackburn JT, Harkey MS, Creighton RA, Kamath GM, Healy K, Schmitz R, Driban JB, Marshall SW, Jordan JM, Spang JT. Associations between cartilage proteoglycan density and patient outcomes 12months following anterior cruciate ligament reconstruction. Knee. 2018 Jan;25(1):118-129. doi: 10.1016/j.knee.2017.10.005. Epub 2018 Jan 9. PMID 29329888
- [Background] Freedson PS, Melanson E, Sirard J. Calibration of the Computer Science and Applications, Inc. accelerometer. Med Sci Sports Exerc. 1998 May;30(5):777-81. doi: 10.1097/00005768-199805000-00021. PMID 9588623
- [Background] McClain JJ, Sisson SB, Tudor-Locke C. Actigraph accelerometer interinstrument reliability during free-living in adults. Med Sci Sports Exerc. 2007 Sep;39(9):1509-14. doi: 10.1249/mss.0b013e3180dc9954. PMID 17805082
- [Background] Roos EM, Roos HP, Ekdahl C, Lohmander LS. Knee injury and Osteoarthritis Outcome Score (KOOS)--validation of a Swedish version. Scand J Med Sci Sports. 1998 Dec;8(6):439-48. doi: 10.1111/j.1600-0838.1998.tb00465.x. PMID 9863983
- [Background] Salavati M, Akhbari B, Mohammadi F, Mazaheri M, Khorrami M. Knee injury and Osteoarthritis Outcome Score (KOOS); reliability and validity in competitive athletes after anterior cruciate ligament reconstruction. Osteoarthritis Cartilage. 2011 Apr;19(4):406-10. doi: 10.1016/j.joca.2011.01.010. Epub 2011 Jan 19. PMID 21255667
- [Background] Xu X, Tupy S, Robertson S, Miller AL, Correll D, Tivis R, Nigg CR. Successful adherence and retention to daily monitoring of physical activity: Lessons learned. PLoS One. 2018 Sep 20;13(9):e0199838. doi: 10.1371/journal.pone.0199838. eCollection 2018. PMID 30235221
- [Background] Adams MA, Sallis JF, Norman GJ, Hovell MF, Hekler EB, Perata E. An adaptive physical activity intervention for overweight adults: a randomized controlled trial. PLoS One. 2013 Dec 9;8(12):e82901. doi: 10.1371/journal.pone.0082901. eCollection 2013. PMID 24349392
- [Background] Hurley JC, Hollingshead KE, Todd M, Jarrett CL, Tucker WJ, Angadi SS, Adams MA. The Walking Interventions Through Texting (WalkIT) Trial: Rationale, Design, and Protocol for a Factorial Randomized Controlled Trial of Adaptive Interventions for Overweight and Obese, Inactive Adults. JMIR Res Protoc. 2015 Sep 11;4(3):e108. doi: 10.2196/resprot.4856. PMID 26362511
- [Background] Kuenze C, Lisee C, Pfeiffer KA, Cadmus-Bertram L, Post EG, Biese K, Bell DR. Sex differences in physical activity engagement after ACL reconstruction. Phys Ther Sport. 2019 Jan;35:12-17. doi: 10.1016/j.ptsp.2018.10.016. Epub 2018 Oct 26. PMID 30396146
- [Background] Kuenze C, Cadmus-Bertram L, Pfieffer K, Trigsted S, Cook D, Lisee C, Bell D. Relationship Between Physical Activity and Clinical Outcomes After ACL Reconstruction. J Sport Rehabil. 2019 Feb 1;28(2):180-187. doi: 10.1123/jsr.2017-0186. Epub 2018 Oct 15. PMID 29140161
- [Background] Lisee CM, Montoye AHK, Lewallen NF, Hernandez M, Bell DR, Kuenze CM. Assessment of Free-Living Cadence Using ActiGraph Accelerometers Between Individuals With and Without Anterior Cruciate Ligament Reconstruction. J Athl Train. 2020 Sep 1;55(9):994-1000. doi: 10.4085/1062-6050-425-19. PMID 32818959

RESULTS

PARTICIPANT FLOW:
Groups:
- Physical Activity Promotion Group: Participants will receive a text message each morning with a personalized, daily step count goal and a link used to confirm receipt of the goal. The preceding 10 days of step data will be rank ordered and the 60th percentile step count will be set as the goal for the next day.
  Physical Activity Promotion: After enrolling, participants will be outfitted with a Fitbit Charge 2 activity monitor. The monitor will be worn during all waking hours, and compliance will be considered as a day with ≥ 1,000 steps. Participants will complete a 14-day "run-in" observation period while wearing the Fitbit but no physical activity (PA) promotion will occur. Individuals who are noncompliant during the "run in" period (<10 days with <1,000 steps) will be removed. Participants will receive a text message each morning with a personalized, daily step count goal and a link used to confirm receipt of the goal. The preceding 10 days of step data will be rank ordered and the 60th percentile step count will be set as the goal for the next day.
Period: Overall Study
Arm/Group | Physical Activity Promotion Group
Started | 7
Completed | 6
Not Completed | 1
Not completed — Lack of time | 1

BASELINE CHARACTERISTICS:
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.7 (5.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: T1rho Relaxation Times in the Medial Femoral Condyle at Baseline
Description: MRI marker of T1rho relaxation times of medial femoral articular cartilage (i.e proteoglycan density) at pre-intervention (baseline)
Time Frame: pre-intervention (baseline)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 53.48 (4.58)

2. Primary Outcome: T1rho Relaxation Times in the Medial Femoral Condyle Post-intervention
Description: MRI marker of T1rho relaxation times of medial femoral articular cartilage (i.e proteoglycan density) at post-intervention (~8 weeks)
Time Frame: post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 52.98 (3.23)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Cohen's d effect size = 0.13, 95% CI 2-sided [-0.68 to 0.93]

3. Primary Outcome: T1rho Relaxation Times in the Lateral Femoral Condyle at Baseline
Description: MRI marker of T1rho relaxation times of lateral femoral articular cartilage (i.e., proteoglycan density) at pre-intervention (baseline)
Time Frame: pre-intervention (baseline)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 51.40 (2.69)

4. Primary Outcome: T1rho Relaxation Times in the Lateral Femoral Condyle Post-intervention
Description: MRI marker of T1rho relaxation times of lateral femoral articular cartilage (i.e proteoglycan density) at post-intervention (~8 weeks)
Time Frame: post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 50.60 (2.48)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Cohen's d effect size = 0.42, 95% CI 2-sided [-0.44 to 1.24]

5. Primary Outcome: T1rho Relaxation Times in the Medial Tibial Condyle at Baseline
Description: MRI marker of T1rho relaxation times of medial tibial articular cartilage (i.e proteoglycan density) at pre-intervention (baseline)
Time Frame: pre-intervention (baseline)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 54.48 (3.62)

6. Primary Outcome: T1rho Relaxation Times in the Medial Tibial Condyle Post-intervention
Description: MRI marker of T1rho relaxation times of medial tibial articular cartilage (i.e proteoglycan density) at post-intervention (~8 weeks)
Time Frame: post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 53.38 (3.03)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Cohen's d effect size = 0.85, 95% CI 2-sided [-0.13 to 1.77]

7. Primary Outcome: T1rho Relaxation Times in the Lateral Tibial Condyle at Baseline
Description: MRI marker of T1rho relaxation times of lateral tibial articular cartilage (i.e proteoglycan density) at pre-intervention (baseline)
Time Frame: pre-intervention (baseline)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 51.69 (4.92)

8. Primary Outcome: T1rho Relaxation Times in the Lateral Tibial Condyle Post-intervention
Description: MRI marker of T1rho relaxation times of lateral tibial articular cartilage (i.e proteoglycan density) at post-intervention (~8 weeks)
Time Frame: post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | 50.51 (4.36)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Cohen's d effect size = 0.97, 95% CI 2-sided [-0.05 to 1.93]

9. Primary Outcome: Change in Daily Steps
Description: Change in average steps per day over 7 day physical activity monitor wear pre-intervention (baseline) to approximately 8-weeks after physical activity promotion intervention
Time Frame: pre-intervention (baseline), post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: steps/day
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
steps/day | 2054 (3795)

10. Primary Outcome: Change in T1rho Relaxation Times in the Medial Femoral Condyle
Description: Change in MRI marker of T1rho relaxation times of medial femoral articular cartilage (i.e proteoglycan density) from pre-intervention (baseline) to approximately 8-weeks after physical activity promotion intervention
Time Frame: pre-intervention (baseline), post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | -0.50 (3.71)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Pearson's r Correlation Coefficient = 0.32, 95% CI 2-sided [-0.67 to 0.90]

11. Primary Outcome: Change in T1rho Relaxation Times in the Medial Tibial Condyle
Description: Change in MRI marker of T1rho relaxation times of medial tibial articular cartilage (i.e proteoglycan density) from pre-intervention (baseline) to approximately 8-weeks after physical activity promotion intervention
Time Frame: pre-intervention (baseline), post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | -1.11 (1.31)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Pearson's r Correlation Coefficient = 0.55, 95% CI 2-sided [-0.48 to 0.94]

12. Primary Outcome: Change in T1rho Relaxation Times in the Lateral Femoral Condyle
Description: change in MRI marker of T1rho relaxation times of lateral femoral articular cartilage (i.e proteoglycan density) from pre-intervention (baseline) to approximately 8-weeks after physical activity promotion intervention
Time Frame: pre-intervention (baseline), post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | -0.81 (1.91)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Pearson's r Correlation Coefficient = 0.23, 95% CI 2-sided [-0.88 to 0.71]

13. Primary Outcome: Change in T1rho Relaxation Times in the Lateral Tibial Condyle
Description: change in MRI marker of T1rho relaxation times of lateral tibial articular cartilage (i.e proteoglycan density) from pre-intervention (baseline) to approximately 8-weeks after physical activity promotion intervention
Time Frame: pre-intervention (baseline), post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: ms
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
ms | -1.18 (1.22)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Pearson's r Correlation Coefficient = -0.19, 95% CI 2-sided [-0.87 to 0.73]

14. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score Quality of Life Subscale
Description: Knee injury Osteoarthritis Outcome Score (KOOS) Quality of Life subscale to measure knee-related quality of life at pre-intervention (baseline). A higher score indicates better knee-related quality of life. Min = 0 and Max = 100
Time Frame: pre-intervention (baseline)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
score on a scale | 63.5 (22.5)

15. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score Quality of Life Subscale
Description: Knee injury Osteoarthritis Outcome Score Quality of Life subscale (KOOS) Quality of Life subscale to measure knee-related quality of life at post-intervention. A higher score indicates better knee-related quality of life. Min = 0 and Max = 100
Time Frame: post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
score on a scale | 69.8 (25.4)
Statistical Analysis 1: Comparison: Physical Activity Promotion Group; Test type: Other; Cohen's d effect size = -0.42, 95% CI 2-sided [-1.24 to 0.44]

16. Other Pre Specified Outcome: Percentage of Patients Retained at Post-intervention Visit (~8 Weeks) Physical Activity Promotion Intervention Retention
Description: physical activity promotion intervention retention
Time Frame: post-intervention (~8 weeks)
Measure: Number; unit: percentage of participants
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 7
percentage of participants | 86

17. Other Pre Specified Outcome: Percentage of Days Participant is Compliant With Fitbit Monitor Wear (>1,000 Steps Per Day)
Description: physical activity promotion intervention compliance
Time Frame: up to post-intervention (~8 weeks)
Measure: Mean (Standard Deviation); unit: percent of days
Arm/Group | Physical Activity Promotion Group
Number analyzed (Participants) | 6
percent of days | 98.00 (0.02)

ADVERSE EVENTS:
Time Frame: From the time of signing informed consent through the Follow-up visit, a total of approximately 3 months.
Arm/Group | Physical Activity Promotion Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-26): https://cdn.clinicaltrials.gov/large-docs/99/NCT04906499/Prot_SAP_001.pdf
  • Informed Consent Form (2022-05-02): https://cdn.clinicaltrials.gov/large-docs/99/NCT04906499/ICF_000.pdf